CLINICAL TRIAL: NCT04604119
Title: Anxiety and Burnout in Anesthetists and Intensive Care Unit Nurses During Covid-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sultan Acar Sevinç, medical doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 1577
Record Dates: First submitted 2020-10-25; First posted 2020-10-27 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Sars-CoV2; Anxiety; Burnout
Keywords: anxiety; burnout; covid 19
MeSH Terms: conditions — Anxiety Disorders; Burnout, Psychological; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim is to measure anxiety level and burnout frequency of healthcare workers including attending physicians, residents and nurses working at intensive care unit during COVID-19 pandemic.

The study protocol had consisted of three parts. The first part was related to demographic details including age, sex, marital status, working position, past medical history.

The second part of the survey was validated Turkish form of Beck anxiety inventory (BAI) It has 21 questions. Every question is a somatic symptom of anxiety. Participants scored them regarding how this symptom bothered them past week. Items have four possible answers: not at all (0 point), mildly (1 point), moderate (2 point), severe (3 point). Total anxiety score can be between 0 and 63. Participants were categorized as no or mild anxiety if the total beck anxiety score was between 0-16, and moderate to severe anxiety if it was more than 16 The last part of the survey was validated Turkish form of Maslach Burnout Inventory (MBI) to evaluate components of BOS

DETAILED DESCRIPTION:
Our institution's ICU has served 31 beds for COVID-19 and 21 beds for other patients during pandemic with 27 attending physicians and 35 residents. Number of night shifts for attending physicians and residents were 3 and 8 per month, respectively. The aim of the study was to evaluate the by measuring anxiety level and burnout frequency of HCWs including attending physicians, residents and nurses in our institution's ICU.

ELIGIBILITY:
Inclusion Criteria:

Healthcare workers in our institute's intensive care units

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Attending physicians, resident doctors, nurses working tertiary intensive care units of our institution
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Anxiety | 10-25 may
  Measured by Beck anxiety inventory. Total anxiety score can be between 0 and 63. Participants were categorized as no or mild anxiety if the total beck anxiety score was between 0-16, and moderate to severe anxiety if it was more than 16

SECONDARY OUTCOMES:
Burnout | 10-25 may
  Measured by Maslach Burnout Inventory. MBI has 7-point 22 Likerd type questions and subdivided into three parts to measure emotional exhaustion (EE) (9 items), depersonalization (DP) (5 items), personal accomplishment (PA) (8 items). High scores on EE and DP subscales and low score on PA subscale imply higher level of burnout

CONTACTS AND LOCATIONS:
Locations (1):
- Sisli Hamidiye Etfal Education and Training Hospital, Istanbul, Turkey (Türkiye)